CLINICAL TRIAL: NCT07299669
Title: The Effect of Bio-electromagnetic-energy-regulation Therapy (BEMER) on Sleep, Readiness to Play and Injuries in Elite Athletes - a Triple Blinded Randomized Controlled Trial
Brief Title: Effects of BEMER Electromagnetic Field Intervention on Sleep, Readiness to Play and Injuries in Elite Athletes
Acronym: BEMER-sport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Western Norway University of Applied Sciences (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ståle Pallesen, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BeSCN 25/1
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Fatigue Recovery
Keywords: BEMER; Athletes; Recovery; Sleep; Injury; Readiness to play; Rate of perceived exertion
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The two arms/conditions involves an electromagnetic mattress and an sham-mattress
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEMER electromagnetic-energy-regulation therapy (Experimental): BEMER electromagnetic mattress; week 1-4 at low lever, week 5-6 medium level and week 7-10 high level
  Interventions: Device: BEMER electromagnetic-energy-regulation therapy
- Sham-mattress (Sham Comparator): Mattress and interface panel similar to the experimental intervention, but without any electromagnetic output signals
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: BEMER electromagnetic-energy-regulation therapy — The BEMER is bio-electric-magnetics-energy-regulation therapy uses a specific waveform of pulsed electromagnetic field (PEMF) to improve microcirculation by 30%. In the present study the bio-electric-magnetics-energy-regulation therapy will be provided through mattresses
  Other Names: BEMER
  Arms: BEMER electromagnetic-energy-regulation therapy
Device: Sham (No Treatment) — Sham mattress with no electromagnetic output
  Arms: Sham-mattress

SUMMARY:
Elite athletes (female football players) will be randomized to 1 of 2 conditions, comprising a BEMER electromagnet field mattress and a sham-mattress. The mattress is to be used in bed for 8 minutes each morning, and for 8 minutes each evening, for 10 weeks. The system has 3 intensity levels - low, medium, and high. The low level will be used for the 4 first weeks, the medium level for the following 2 weeks, and the high level for the last 4 weeks. Those in the sham conditions have a display and mattress looking identical, and follow the same procedure as those in BEMER electromagnet field mattress condition. The primary outcome comprises total sleep time and sleep efficacy assessed with a sleep radar as well as readiness to play (composite measure of daily self-report of fatigue, sleep quality, muscle soreness, stress and mood). Secondary outcomes comprise duration of deep sleep also assessed with the sleep radar, injury severity, and rate of perceived exertion following training and matches. Baseline registrations are conducted for 4 weeks prior to the intervention and outcomes are registered during the last 4 weeks of the intervention.

DETAILED DESCRIPTION:
Contrary to common assumptions, athletes often experience insufficient sleep, particularly in the context of competitive events. Furthermore, a significant proportion of athletes report poor sleep quality, potentially linked to frequent travel, intense training, suboptimal training times and inadequate caloric intake. Female athletes are especially susceptible, facing additional challenges such as role conflicts, gender discrimination, body image concerns, increased risk of eating disturbances, and negative impact from menstruation, all of which may hinder restitution. A promising intervention to enhance and facilitate restitution involves the use of low frequency pulsed electromagnetic field (PEMF) therapy, which has demonstrated the potential to increase blood flow, particularly in micro vessels, and is as such assumed to increase micro-circulation, among other in the skeleton muscles. The effectiveness of PEMF therapy in athletes has so far not been investigated using a randomized controlled design.

In this study, a triple blind (participants, researchers and statistician) randomized controlled trial will be undertaken, with female athletes (N=60) from national (Norway) football teams being randomly designed to receive either a placebo mattress or a PEMF-mattress based on a 1:1 ratio, using stratified randomization by team. During a baseline assessment period of 4 weeks, 3 primary outcomes (radar assessed total sleep time and sleep efficiency), and readiness to play (composite measure of daily self-report of fatigue, sleep quality, muscle soreness, stress and mood) will be recorded at a daily basis. These 3 outcomes will be analyzed also specifically for the day/night following matches (as secondary outcomes). Other secondary outcomes comprise the amount (duration) of slow wave sleep/deep, assessed with the sleep radar technology, the severity of injuries, and the rate of perceived exertion (RPE) following training and matches.

The participants (N=60) will following the 4-week baseline registration commence a 10 week intervention phase involving daily use of the mattress for 2 (morning and evening) x 8 minutes. The system has 3 levels of PEMF-intensity (low, medium, high). The first four weeks the low intensity will be used, the next two the medium intensity will be used, thereafter (last four weeks) the high intensity will be used. This intervention period will be accompanied by reassessment of the primary and secondary outcomes during the last 4 weeks of the 10-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Female elite football player in Norway
* Playing on team willing to part-take in the study

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Total sleep time | Change from baseline (4 weeks before interventions) to the last 4 weeks of the intervention.
  Total sleep time in the main sleep episode assessed with the sleep radar Somnofy, expressed as minutes per day. High total sleep time is regarded as a more positive outcome than a lower total sleep time.
Sleep efficiency | Change from baseline (4 weeks before intervention) to the last 4 weeks of the intervention
  Percentage of time in bed following shut-eye (lights out) to rising from bed where the participant did sleep - assessed with the sleep radar Somnofy during the main sleep period. The measure comprises the percentage of time being asleep, and higher values (percentage) are regarded as a better outcome than lower values (percentage).
Readiness to play | Change from baseline (4 weeks before intervention) to the last 4 weeks of the intervention
  Daily morning self-report on an adapted version of the Hooper Index (Hooper, Mackinnon, Howard, Gordon, & Bachmann, 1995), comprising four items assessing fatigue, sleep quality, muscle soreness, and stress. Each item is rated on a 7-point scale ranging from 1 to 7 (where 7 is the worst state and 1 is the best state). A composite daily score ranging from 4 to 28 is calculated - lower scores are associated with the best outcomes.

SECONDARY OUTCOMES:
Total sleep time the day following matches | Change from baseline (4 weeks before interventions) to the last 4 weeks of the intervention exclusively on the nights after matches.
  Total sleep time in the main sleep episode assessed with the sleep radar Somnofy the day following matches, expressed as minutes per day. High total sleep time is regarded as a more positive outcome than a lower total sleep time.
Sleep efficiency the day following matches | Change from baseline (4 weeks before intervention) to the last 4 weeks of the intervention exclusively the night following matches.
  Percentage of time in bed following shut-eye (lights out) to rising from bed where the participant did sleep assessed with the sleep radar Somnofy during the main sleep period - the day following matches. The measure comprises the percentage of time being asleep, and higher values (percentage) are regarded as a better outcome than lower values (percentage).
Readiness to play the day after matches | Change from baseline (4 weeks before intervention) to the last 4 weeks of the intervention, exclusively on the day after matches.
  Daily morning self-report on an adapted version of the Hooper Index (Hooper, Mackinnon, Howard, Gordon, & Bachmann, 1995), comprising four items assessing fatigue, sleep quality, muscle soreness, and stress. Each item is rated on a 7-point scale ranging from 1 to 7 (where 7 is the worst state and 1 is the best state). A composite daily score ranging from 4 to 28 is calculated - lower scores are associated with the best outcomes.
Deep sleep duration | Change from baseline (4 weeks before intervention) to the last 4 weeks of the intervention
  Deep sleep duration assessed with the sleep radar Somnofy during the main sleep period, expressed in minutes. Higher values are regarded as better outcomes than lower values
Health problems | Change from baseline (4 weeks before interventions) to the last 4 weeks of the intervention.
  Health problems are assessed with the Oslo Sports Trauma Research Center Questionnaire on Health Problems-2. The questionnaire has four items (degree of health problem impact on: 1) participation in training, 2) modification of training, 3) performance, and 4) pain). All items have four response alternatives and each is scored 0-8-17-25. A composite score ranging from 0-100 is calculated - higher numbers reflect higher health problem severity. The instrument will be administered once per week.
Rate of perceived exertion | Change from baseline (4 weeks before interventions) to the last 4 weeks of the intervention.
  Rate of Perceived Exertion (RPE) following training and matches as measured by a single item based on the Borg CR-10 scale (Borg, 1990). The response alternatives ranges from 0 (no exertion) to 10 (maximal exertion). Lower values are regarded as better outcomes than higher values.

CONTACTS AND LOCATIONS:
Overall Officials: Ståle Pallesen, PhD, Principal Investigator — University of Bergen
Locations (2):
- Norway (2):
  - Bergensregionen, Bergen
  - Osloregionen, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Complete dataset
Supporting Information: Study Protocol
Time Frame: From January 1, 2027
Access Criteria: Researchers with a phd and relevant background can access the material. In order to get the material they need to contact the PI. They will be provided with the study protocol